CLINICAL TRIAL: NCT05028569
Title: Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study of BOTOX (Botulinum Toxin Type A) for the Prevention of Migraine in Subjects With Episodic Migraine
Brief Title: Study of BOTOX Injections in Prevention of Migraine in Adult Participants With Episodic Migraine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to lack of efficacy from the primary analysis results.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M21-307; 2021-001979-16 (EudraCT Number)
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Episodic Migraine
Keywords: Migraine; Episodic Migraine; BOTOX; Botulinum Toxin Type A
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Double-Blind Phase: Placebo (Placebo Comparator): Participants received placebo for BOTOX intramuscular injections in the head/neck muscles on Day 1 and Week 12.
  Interventions: Drug: Placebo
- Double-Blind Phase: BOTOX 155 U (Experimental): Participants received intramuscular injections of BOTOX 155 U in the head/neck muscles on Day 1 and Week 12.
  Interventions: Drug: BOTOX
- Double-Blind Phase: BOTOX 195 U (Experimental): Participants received intramuscular injections of BOTOX 195 U in the head/neck muscles on Day 1 and Week 12.
  Interventions: Drug: BOTOX
- Open-Label Phase: BOTOX 195 U (Experimental): Eligible participants received intramuscular injections of BOTOX 195 U in the head/neck muscles on Weeks 24 and 36.
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — Intramuscular Injection
  Other Names: Botulinum Toxin Type A
  Arms: Double-Blind Phase: BOTOX 155 U; Double-Blind Phase: BOTOX 195 U; Open-Label Phase: BOTOX 195 U
Drug: Placebo — Intramuscular Injection
  Arms: Double-Blind Phase: Placebo

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound (International Classification of Headache Disorders, 2018). Migraine can be further categorized according to the frequency of attacks as episodic migraine (EM) or chronic migraine (CM). This study will assess the effects of BOTOX in preventing migraine in adult participants with EM.

BOTOX is being developed for the prevention of migraine in adults with episodic migraine (EM). Participants will be enrolled in 3 different treatment groups. There is 1 in 3 chance that participants will be assigned to receive placebo. Approximately 777 adult participants with EM will be enrolled in approximately 125 sites across the world.

Participants will receive intramuscular injections (injected into the muscle) of BOTOX or Placebo on Day 1 and Week 12. Eligible participants will receive BOTOX on Week 24 and Week 36.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine headache disorder meeting International Classification of Headache Disorders (ICHD)-3 diagnostic criteria for migraine with aura or migraine without aura for >= 12 months.
* Onset of migraine before 50 years of age.
* History of 6 to 14 migraine days/month in each of the 3 months prior to Visit 1.
* Six to 14 migraine/probable migraine days during the 4-week screening/baseline phase.
* Less than 15 headache days/month in each of the 3 months prior to Visit 1 and during the 4-week screening/baseline phase.

Exclusion Criteria:

* Current diagnosis of chronic migraine according to ICHD-3.
* History or current diagnosis of migraine with brainstem aura, retinal migraine, complications of migraine, chronic tension-type headache, trigeminal autonomic cephalalgias, hypnic headache, hemicrania continua, or new daily persistent headache.
* History of headache attributed to another disorder (e.g., cervical dystonia, craniotomy, head/neck trauma) with exception that medication overuse headache per ICHD-3 criteria is allowed.
* History of inadequate response to > 4 prophylactic treatment for migraine, 2 of which have different mechanisms of action.
* Female who is pregnant, breastfeeding, or considering becoming pregnant during the study or within 90 days after the last dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (133):
- United States (82):
  - Neurology and Neurodiagnostics of Alabama /ID# 231918, Hoover, Alabama
  - Rehabilitation & Neurological Services /ID# 252441, Huntsville, Alabama
  - Alea Research /ID# 233329, Phoenix, Arizona
  - Duplicate_Barrow Neurological Institute /ID# 231799, Phoenix, Arizona
  - Clinical Endpoints /ID# 232625, Scottsdale, Arizona
  - Tucson Neuroscience Research /ID# 232288, Tucson, Arizona
  - Arkansas Clinical Research /ID# 231640, Little Rock, Arkansas
  - Woodland International Research Group /ID# 231492, Little Rock, Arkansas
  - Hope Clinical Research /ID# 232189, Canoga Park, California
  - Pharmacology Research Institute (PRI) - Encino (Wake) /ID# 231351, Encino, California
  - Duplicate_Neuro Pain Medical Center /ID# 231478, Fresno, California
  - Sun Valley Research Center /ID# 231350, Imperial, California
  - Wake Research - Pharmacology Research Institute (WR-PRI), LLC (Alamitos) /ID# 231908, Los Alamitos, California
  - Pharmacology Research Institute (PRI) - Newport Beach (Wake) /ID# 231337, Newport Beach, California
  - Colorado Springs Neurological Associates (CSNA) /ID# 230662, Colorado Springs, Colorado
  - Summit Headache and Neurologic Institute /ID# 231809, Englewood, Colorado
  - Advanced Neurosciences Research, LLC /ID# 230658, Fort Collins, Colorado
  - Georgetown University Hospital /ID# 232129, Washington D.C., District of Columbia
  - Neurology Offices of South Florida, PLLC /ID# 232281, Boca Raton, Florida
  - Nova Clinical Research, LLC /ID# 245256, Bradenton, Florida
  - Velocity Clinical Research - Hallandale Beach /ID# 232442, Hallandale, Florida
  - CNS Healthcare - Jacksonville /ID# 231345, Jacksonville, Florida
  - Brainstorm Research /ID# 243825, Miami, Florida
  - Sensible Healthcare /ID# 231340, Ocoee, Florida
  - Clinical Neuroscience Solutions, Inc /ID# 231362, Orlando, Florida
  - Pain Relief Centers /ID# 232415, Sun City Center, Florida
  - University of South Florida- Neuroscience Institute /ID# 231808, Tampa, Florida
  - Olympian Clinical Research - Tampa /ID# 239519, Tampa, Florida
  - Accel Research Sites - Tampa Clinical Research Unit /ID# 231670, Tampa, Florida
  - Premiere Research Institute - Palm Beach /ID# 230646, West Palm Beach, Florida
  - Conquest Research /ID# 232604, Winter Park, Florida
  - Accel Research Sites Neurostudies /ID# 230665, Decatur, Georgia
  - CenExcel iResearch LLC /ID# 231335, Decatur, Georgia
  - Clinical Research Institute /ID# 239517, Stockbridge, Georgia
  - Northwest Clinical Trials /ID# 230657, Boise, Idaho
  - Velocity Clinical Research - Boise /ID# 230660, Meridian, Idaho
  - Robbins Headache Clinic /ID# 230970, Riverwoods, Illinois
  - Josephson-Wallack-Munshower Neurology - Northeast /ID# 230654, Indianapolis, Indiana
  - Deaconess Clinic - Gateway Health Center /ID# 231329, Newburgh, Indiana
  - Duplicate_Accellacare - McFarland Clinic /ID# 231496, Ames, Iowa
  - Kansas Institute of Research /ID# 231862, Overland Park, Kansas
  - Ochsner Clinic Foundation /ID# 230645, Covington, Louisiana
  - Brigham and Women's Faulkner Hospital /ID# 231865, Boston, Massachusetts
  - Boston Clinical Trials /ID# 231367, Boston, Massachusetts
  - Michigan Headache & Neurological Institute (MHNI) /ID# 230659, Ann Arbor, Michigan
  - Minneapolis Clinic of Neurology - Burnsville /ID# 231780, Burnsville, Minnesota
  - StudyMetrix Research /ID# 230642, City of Saint Peters, Missouri
  - Clinvest Research LLC /ID# 252440, Springfield, Missouri
  - Excel Clinical Research /ID# 232188, Las Vegas, Nevada
  - Las Vegas Clinical Trials /ID# 232628, North Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc. /ID# 231101, Albuquerque, New Mexico
  - Duplicate_Dent Neurosciences Research Center, Inc. /ID# 252442, Amherst, New York
  - Fieve Clinical Research, Inc. /ID# 231365, New York, New York
  - Montefiore Headache Center /ID# 232130, The Bronx, New York
  - Upstate Clinical Research Associates /ID# 231343, Williamsville, New York
  - Headache Wellness Center /ID# 230819, Greensboro, North Carolina
  - M3 Wake Research Inc. /ID# 232285, Raleigh, North Carolina
  - Neurology - Triad /ID# 231733, Winston-Salem, North Carolina
  - Duplicate_Duplicate_University Of Cincinnati Medical Center /ID# 231739, Cincinnati, Ohio
  - IPS Research Company /ID# 231085, Oklahoma City, Oklahoma
  - Lynn Institute of Oklahoma City /ID# 231349, Oklahoma City, Oklahoma
  - Cutting Edge Research Group /ID# 231095, Oklahoma City, Oklahoma
  - Sooner Clinical Research /ID# 231096, Oklahoma City, Oklahoma
  - Abington Neurological Associates - Abington /ID# 231798, Abington, Pennsylvania
  - Lehigh Center for Clinical Research /ID# 231355, Allentown, Pennsylvania
  - Suburban Research Associates - Media /ID# 231354, Media, Pennsylvania
  - Jefferson Hospital for Neuroscience /ID# 230664, Philadelphia, Pennsylvania
  - Duplicate_Frontier Clinical Research /ID# 232623, Smithfield, Pennsylvania
  - Clinical Trials of SC /ID# 231369, Charleston, South Carolina
  - Coastal Carolina Research Center - North Charleston /ID# 231353, North Charleston, South Carolina
  - Clinical Neuroscience Solutions - Memphis /ID# 231328, Memphis, Tennessee
  - Nashville Neuroscience Group /ID# 231642, Nashville, Tennessee
  - Austin Clinical Trial Partners /ID# 231092, Austin, Texas
  - Texas Neurology /ID# 230661, Dallas, Texas
  - NeuroCare Plus /ID# 252499, Houston, Texas
  - Charlottesville Medical Research /ID# 231368, Charlottesville, Virginia
  - Integrated Neurology Services - Falls Church /ID# 244776, Falls Church, Virginia
  - Tidewater Integr Med Research /ID# 231359, Virginia Beach, Virginia
  - Sentara Neurology Specialists - Virginia Beach /ID# 231341, Virginia Beach, Virginia
  - Northwest Clinical Research Center /ID# 231336, Bellevue, Washington
  - Puget Sound Neurology /ID# 230640, Tacoma, Washington
  - Frontier Clinical Research - Kingwood /ID# 234127, Kingwood, West Virginia
- Canada (5):
  - CHAMP Clinic /ID# 231635, Calgary, Alberta
  - Vancouver Island Health Authority /ID# 231992, Victoria, British Columbia
  - Maritime Neurology /ID# 232048, Halifax, Nova Scotia
  - Toronto Memory Program /ID# 240006, Toronto, Ontario
  - Clinique Neuro Levis /ID# 232049, Lévis, Quebec
- Czechia (7):
  - Fakultní Nemocnice U Sv. Anny V Brně /ID# 232213, Brno, Brno-mesto
  - Fakultni Nemocnice Ostrava /ID# 232211, Ostrava, Ostrava-mesto
  - Nemocnice Jihlava, prispevkova organizace /ID# 232164, Jihlava
  - Clintrial s.r.o. /ID# 232208, Prague
  - DADO MEDICAL s.r.o. /ID# 232157, Prague
  - Axon Clinical, s.r.o. /ID# 232212, Prague
  - Fakultni Thomayerova nemocnice /ID# 232214, Prague
- Germany (10):
  - Duplicate_Neurologie Klinikum Großhadern /ID# 232479, Munich, Bavaria
  - Duplicate_Kopfschmerzzentrum Frankfurt /ID# 234066, Frankfurt am Main, Hesse
  - Universitaetsmedizin Rostock /ID# 232471, Rostock, Mecklenburg-Vorpommern
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 239283, Dresden, Saxony
  - Schmerzklinik Kiel /ID# 232480, Kiel, Schleswig-Holstein
  - Zentrum für Neurologie, Neurochirurgie und Psychiatrie /ID# 232472, Berlin
  - Praxis Dr. Gendolla /ID# 232474, Essen
  - Universitaetsklinikum Essen /ID# 232478, Essen
  - Universitaetsklinikum Halle (Saale) /ID# 241506, Halle
  - Vitos Orthopaedische Klinik Kassel gemeinnuetzige GmbH /ID# 232475, Kassel
- Israel (6):
  - Maccabi Healthcare Services /ID# 238605, Kfar Saba, Central District
  - Hillel Yaffe Medical Center /ID# 232122, Hadera, Haifa District
  - Shaare Zedek Medical Center /ID# 239485, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 232119, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 232598, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 238732, Haifa
- Poland (8):
  - Solumed Centrum Medyczne /ID# 238446, Poznan, Greater Poland Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o. /ID# 233526, Krakow, Lesser Poland Voivodeship
  - Linden Sp. z o.o. sp.k. /ID# 245685, Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia Dr Boczarska Jedynak /ID# 251857, Oświęcim, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 232355, Lublin, Lublin Voivodeship
  - Warszawska Klinika Sp. z o.o. /ID# 240612, Warsaw, Masovian Voivodeship
  - Silmedic Sp. z o.o. /ID# 232358, Katowice, Silesian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak /ID# 241887, Wroclaw
- Spain (6):
  - Clinica Universidad de Navarra - Pamplona /ID# 232270, Pamplona, Navarre
  - Hospital Universitario Central de Asturias /ID# 232428, Oviedo, Principality of Asturias
  - Hospital Universitario Vall d'Hebron /ID# 232268, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 233320, Madrid
  - Hospital Universitario La Paz /ID# 232495, Madrid
  - Hospital Clinico Universitario de Valladolid /ID# 232272, Valladolid
- Sweden (4):
  - Skaneuro Privatmottagning /ID# 232175, Lund, Skåne County
  - Neurology Clinic /ID# 234067, Stockholm, Stockholm County
  - Optimuskliniken /ID# 232174, Upplands Vasby
  - Linkoping University Hospital /ID# 234040, Linköping, Östergötland County
- United Kingdom (5):
  - Hull University Teaching Hospitals NHS Trust /ID# 242763, Hull, East Riding Of Yorkshire
  - Duplicate_Queen Elizabeth University Hospital /ID# 244870, Glasgow, Glasgow City
  - NHS Highland /ID# 242855, Inverness
  - Walton Centre /ID# 242857, Liverpool
  - St Pancras Clinical Research /ID# 242764, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 118 sites in 9 countries and was initiated in November 2021. Adults with episodic migraine (EM) were eligible.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to receive 2 treatment cycles of BOTOX 195 U, BOTOX 155 U, or placebo. BOTOX (155 U or 195 U) or matching placebo was administered by a trained injector at Day 1 and Week 12 of the Double-Blind Phase. Those who continued to the Open-label Phase received BOTOX 195 U at 12-week intervals for up to 2 treatment cycles.
Groups:
- Screening/Baseline Phase: Participants with 6 to 14 migraine days and < 15 headache days per month in each of the 3 months prior to the screening visit (Visit 1) and during the 4-week Screening/Baseline Phase were randomized in this study.
- Double-Blind Phase: Placebo: Participants randomized to receive placebo intramuscular injections in the head/neck muscles for BOTOX on Day 1 and Week 12.
- Double-Blind Phase: BOTOX 155 U: Participants randomized to receive intramuscular injections in the head/neck muscles of BOTOX 155 U on Day 1 and Week 12.
- Double-Blind Phase: BOTOX 195 U: Participants randomized to receive intramuscular injections in the head/neck muscles of BOTOX 195 U on Day 1 and Week 12.
- Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U: Participants randomized to receive placebo for BOTOX intramuscular injections in the head/neck muscles on Day 1 and Week 12 during the Double-Blind Phase who then received intramuscular injections of BOTOX 195 U in the head/neck muscles on Weeks 24 and 36 in the Open-Label Phase.
- Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U: Participants randomized to receive intramuscular injections of BOTOX 155 U in the head/neck muscles on Day 1 and Week 12 during the Double-Blind Phase who then received intramuscular injections of BOTOX 195 U in the head/neck muscles on Weeks 24 and 36 in the Open-Label Phase.
- Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U: Participants randomized to receive intramuscular injections of BOTOX 195 U in the head/neck muscles on Day 1 and Week 12 during the Double-Blind Phase who then received intramuscular injections of BOTOX 195 U in the head/neck muscles on Weeks 24 and 36 in the Open-Label Phase.
Period: Screening/Baseline Phase
Arm/Group | Screening/Baseline Phase | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U | Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U
Started | 775 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 775 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Phase
Arm/Group | Screening/Baseline Phase | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U | Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U
Started | 0 | 257 | 257 | 261 | 0 | 0 | 0
Received at Least One Dose of Study Treatment | 0 | 257 | 256 | 261 | 0 | 0 | 0
Completed | 0 | 217 | 230 | 223 | 0 | 0 | 0
Not Completed | 0 | 40 | 27 | 38 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 6 | 3 | 9 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 27 | 20 | 22 | 0 | 0 | 0
Not completed — Other, not specified | 0 | 5 | 4 | 6 | 0 | 0 | 0
Period: Open-Label Phase
Arm/Group | Screening/Baseline Phase | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U | Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U
Started | 0 | 0 | 0 | 0 | 217 | 230 | 223
Completed | 0 | 0 | 0 | 0 | 186 | 199 | 192
Not Completed | 0 | 0 | 0 | 0 | 31 | 31 | 31
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 5 | 5 | 4
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 15 | 8 | 13
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 4 | 10 | 5
Not completed — Other, not specified | 0 | 0 | 0 | 0 | 6 | 5 | 7
Not completed — Completed Double-Blind Phase and then withdrew from study | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Completed Double-Blind Phase and then withdrew due to pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (as randomized)
Groups:
- Double-Blind Phase: Placebo: Participants received placebo intramuscular injections in the head/neck muscles for BOTOX on Day 1 and Week 12.
- Double-Blind Phase: BOTOX 155 U: Participants received intramuscular injections in the head/neck muscles of BOTOX 155 U on Day 1 and Week 12.
- Double-Blind Phase: BOTOX 195 U: Participants received intramuscular injections in the head/neck muscles of BOTOX 195 U on Day 1 and Week 12.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U | Total
Number analyzed (Participants) | 257 | 257 | 261 | 775
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.12) | 41.1 (10.37) | 41.1 (10.76) | 40.8 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231 | 227 | 224 | 682
  Male | 26 | 30 | 37 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 30 | 37 | 91
  Not Hispanic or Latino | 233 | 227 | 224 | 684
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 3 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 23 | 12 | 14 | 49
  White | 229 | 240 | 237 | 706
  More than one race | 2 | 0 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Frequency of Monthly Migraine Days Across Months 5 and 6
Description: The frequency of monthly migraine days across Months 5 and 6 is calculated by taking the 2-month average of monthly migraine days over Months 5 and 6. Month 5 and Month 6 are the 28-day daily diary periods ending with Days 56 and Days 84 after the second study treatment intervention day with BOTOX or placebo injections, respectively. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Months 5-6
Population: Intent-to-Treat Population (as Randomized); data used are "observed data" (without imputation for missing values)
Measure: Least Squares Mean (95% Confidence Interval); unit: monthly migraine days
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U
Number analyzed (Participants) | 227 | 234 | 227
monthly migraine days | -3.0 [-3.55 to -2.46] | -3.1 [-3.65 to -2.57] | -3.0 [-3.51 to -2.43]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 195 U; BOTOX 195 U vs Placebo; Test type: Superiority — P-value/95% CI obtained from mixed-effects model for repeated measures (MMRM) for primary analysis of the 2 visits across Months 5 and 6. Tx (BOTOX 195 U, 155 U, placebo), month (Months 1-6), country, strata of previous exposure to migraine prophylactic treatment, and Tx group-by-month interaction as fixed effects, with Baseline monthly migraine days as covariate, included as a continuous variable rather than the binomial stratification variable. Subject/residual errors are random effects; p = 0.914, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.62 to 0.69], Standard Error of Mean 0.33 — LS Mean Difference = BOTOX 195 U - Placebo
Statistical Analysis 2: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 155 U; BOTOX 155 U vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.745, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.1, 95% CI 2-sided [-0.76 to 0.55], Standard Error of Mean 0.33 — LS Mean Difference = BOTOX 155 U - Placebo

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: Double-Blind Phase (Week 0-24); Open-Label Phase (Week 24-48)
Population: Safety Analysis Set: all participants who received any amount of study treatment; included in the analysis according to the study treatment that they actually received (as treated).
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U: Participants who received placebo for BOTOX intramuscular injections in the head/neck muscles on Day 1 and Week 12 during the Double-Blind Phase who then received intramuscular injections of BOTOX 195 U in the head/neck muscles on Weeks 24 and 36 in the Open-Label Phase.
- Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U: Participants who received intramuscular injections of BOTOX 155 U in the head/neck muscles on Day 1 and Week 12 during the Double-Blind Phase who then received intramuscular injections of BOTOX 195 U in the head/neck muscles on Weeks 24 and 36 in the Open-Label Phase.
- Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U: Participants who received intramuscular injections of BOTOX 195 U in the head/neck muscles on Day 1 and Week 12 during the Double-Blind Phase who then received intramuscular injections of BOTOX 195 U in the head/neck muscles on Weeks 24 and 36 in the Open-Label Phase.
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U | Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U
Number analyzed (Participants) | 257 | 255 | 262 | 217 | 225 | 223
Participants
  Any TEAE | 106 | 117 | 120 | 76 | 75 | 80
  TESAE | 6 | 3 | 6 | 2 | 1 | 1

3. Secondary Outcome: Change From Baseline in the Frequency of Monthly Headache Days Across Months 5 and 6
Description: The frequency of monthly headache days across Months 5 and 6 is calculated by taking the 2-month average of monthly headache days over Months 5 and 6. Month 5 and Month 6 are the 28-day daily diary periods ending with Days 56 and Days 84 after the second study treatment intervention day with BOTOX or placebo injections, respectively. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Months 5-6
Population: Intent-to-Treat Population (as Randomized); data used are "observed data" (without imputation for missing values)
Measure: Least Squares Mean (95% Confidence Interval); unit: monthly headache days
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U
Number analyzed (Participants) | 227 | 234 | 227
monthly headache days | -3.2 [-3.77 to -2.59] | -3.1 [-3.71 to -2.54] | -2.9 [-3.46 to -2.29]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 195 U; BOTOX 195 U vs Placebo; Test type: Superiority — P-value/95% CI obtained from mixed-effects model for repeated measures (MMRM) for primary analysis of the 2 visits across Months 5 and 6. Tx (BOTOX 195 U, 155 U, placebo), month (Months 1-6), country, strata of previous exposure to migraine prophylactic treatment, and Tx group-by-month interaction as fixed effects, with Baseline monthly headache days as covariate, included as a continuous variable. Subject/residual errors are random effects; p = 0.414, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.3, 95% CI 2-sided [-0.42 to 1.01], Standard Error of Mean 0.36 — LS Mean Difference = BOTOX 195 U - Placebo
Statistical Analysis 2: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 155 U; BOTOX 155 U vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.889, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.1, 95% CI 2-sided [-0.66 to 0.76], Standard Error of Mean 0.36 — LS Mean Difference = BOTOX 155 U - Placebo

4. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction From Baseline in the Frequency of Monthly Migraine Days Across Months 5 and 6
Description: The frequency of monthly migraine days across Months 5 and 6 is calculated by taking the 2-month average of monthly migraine days over Months 5 and 6. Month 5 and Month 6 are the 28-day daily diary periods ending with Days 56 and Days 84 after the second study treatment intervention day with BOTOX or placebo injections, respectively. The responder status of 50% reduction from Baseline is defined as a participant with at least a 50% reduction from Baseline in the 2-month average of monthly migraine days over Months 5 and 6.
Time Frame: Baseline, Months 5-6
Population: Intent-to-Treat Population (as Randomized); data used are "observed data" (without imputation for missing values)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U
Number analyzed (Participants) | 227 | 234 | 227
percentage of participants | 44.9 [38.35 to 51.66] | 46.2 [39.64 to 52.77] | 47.1 [40.50 to 53.85]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 195 U; BOTOX 195 U vs Placebo; Test type: Superiority — P-value is obtained from Logistic Regression. Model includes treatment (BOTOX 195 U, BOTOX 155 U, and placebo), country and strata of previous exposure to migraine prophylactic treatment as fixed effects, with the Baseline monthly migraine days as a covariate, included as a continuous variable. Subject and residual errors are random effects in this by visit logistic covariate analysis of variance (ANCOVA). Confidence intervals (Clopper-Pearson) are based on binomial-distribution assumptions; p = 0.451, Regression, Logistic; Response Rate Difference = 2.2, 95% CI 2-sided [-7.08 to 11.46] — Response Rate Difference = BOTOX 195 U - Placebo
Statistical Analysis 2: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 155 U; BOTOX 155 U vs Placebo; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.762, Regression, Logistic; Response Rate Difference = 1.2, 95% CI 2-sided [-7.94 to 10.40] — Response Rate Difference = BOTOX 155 U - Placebo

5. Secondary Outcome: Change From Baseline in the Frequency of Monthly Acute Headache Medication Days Across Months 5 and 6
Description: Monthly acute headache medication days across Months 5 and 6 is calculated by taking the 2-month average of monthly acute headache medication days over Months 5 and 6. Month 5 and Month 6 are the 28-day daily diary periods ending with Days 56 and Days 84 after the second study treatment intervention day with BOTOX or placebo injections, respectively. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Months 5-6
Population: Intent-to-Treat Population (as Randomized); data used are "observed data" (without imputation for missing values)
Measure: Least Squares Mean (95% Confidence Interval); unit: Monthly Acute Headache Medication Days
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U
Number analyzed (Participants) | 227 | 234 | 227
Monthly Acute Headache Medication Days | -2.0 [-2.47 to -1.47] | -1.9 [-2.44 to -1.44] | -1.8 [-2.34 to -1.35]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 195 U; BOTOX 195 U vs Placebo; Test type: Superiority — P-value/95% CI obtained from mixed-effects model for repeated measures (MMRM) for primary analysis of the 2 visits across Months 5 and 6. Tx (BOTOX 195 U, BOTOX 155 U, placebo), month (Months 1-6), country, strata of previous exposure to migraine prophylactic treatment, and Tx group-by-month interaction as fixed effects, with the Baseline monthly acute headache medication days as a covariate, included as a continuous variable. Subject and residual errors are random effects; p = 0.686, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.1, 95% CI 2-sided [-0.48 to 0.74], Standard Error of Mean 0.31 — LS Mean Difference = BOTOX 195 U - Placebo
Statistical Analysis 2: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 155 U; BOTOX 155 U vs Placebo; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.913, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.57 to 0.64], Standard Error of Mean 0.31 — LS Mean Difference = BOTOX 155 U - Placebo

6. Secondary Outcome: Change From Baseline in Migraine-Specific Quality of Life Questionnaire Version 2.1 (MSQ v2.1) Role Function - Restrictive (RFR) Domain Score At Month 6
Description: The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality of life impairments attributed to migraine over the past 4 weeks. It is divided into 3 domains, and the Role Function Restrictive (RFR) assesses how migraines limit one's daily social and work-related activities using a 6-point scale ranging from "none of the time" to "all of the time". Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores indicate better quality of life. Positive changes from Baseline indicate improvement.
Time Frame: Baseline, Month 6
Population: Intent-to-Treat Population (as Randomized); data used are "observed data" (without imputation for missing values)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U
Number analyzed (Participants) | 216 | 228 | 218
units on a scale | 18.6 [15.77 to 21.51] | 19.4 [16.58 to 22.27] | 19.0 [16.15 to 21.87]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 195 U; BOTOX 195 U vs Placebo; Test type: Superiority — P-value/95% CI obtained from mixed-effects model for repeated measures (MMRM) for primary analysis of the visit at Month 6. Tx (BOTOX 195 U, BOTOX 155 U, placebo), month (Months 1-6), country, strata of previous exposure to migraine prophylactic treatment, and Tx group-by-month interaction as fixed effects, with the Baseline MSQ v2.1 RFR Domain Score as a covariate, included as a continuous variable. Subject and residual errors are random effects; p = 0.837, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.4, 95% CI 2-sided [-3.18 to 3.93], Standard Error of Mean 1.81 — LS Mean Difference = BOTOX 195 U - Placebo
Statistical Analysis 2: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 155 U; BOTOX 155 U vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.662, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.8, 95% CI 2-sided [-2.74 to 4.31], Standard Error of Mean 1.79 — LS Mean Difference = BOTOX 155 U - Placebo

7. Secondary Outcome: Change From Baseline in the Activity Impairment in Migraine - Diary (AIM-D) Physical Impairment Domain Score Across Months 5 and 6
Description: AIM-D Physical Impairment Domain score is calculated based on the summation of AIM-D items 6-9. Participants answer each question based on the level of difficulty experienced in the 24 hours prior, with "during your headache" indicated for when they reported a headache, using a 6-point rating scale ranging from "not difficult at all" to "extremely difficult". The raw daily score is transformed to a 0-100 scale, and the monthly score is calculated using the average daily scores, where a higher score indicates worse physical impairment. AIM-D Physical Impairment domain score across Months 5 and 6 is calculated by taking the 2-month average of AIM-D Physical Impairment domain scores over Months 5 and 6. Month 5 and Month 6 are the 28-day daily diary periods ending with Days 56 and Days 84 after the second study treatment intervention day with BOTOX or placebo injections, respectively. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Months 5-6
Population: Intent-to-Treat Population (as Randomized); data used are "observed data" (without imputation for missing values)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U
Number analyzed (Participants) | 225 | 232 | 222
units on a scale | -5.0 [-6.23 to -3.82] | -4.6 [-5.82 to -3.39] | -4.9 [-6.07 to -3.66]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 195 U; BOTOX 195 U vs Placebo; Test type: Superiority — P-value/95% CI are obtained from mixed-effects model for repeated measures (MMRM) analysis for primary analysis of the 2 visits across Months 5 and 6. Tx (BOTOX 195 U, BOTOX 155 U, placebo), month (Months 1-6), country, strata of previous exposure to migraine prophylactic treatment, and Tx group-by-month interaction as fixed effects, with the Baseline AIM-D Physical Impairment domain score as a covariate, included as a continuous variable. Subject and residual errors are random effects; p = 0.834, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.2, 95% CI 2-sided [-1.32 to 1.63], Standard Error of Mean 0.75 — LS Mean Difference = BOTOX 195 U - Placebo
Statistical Analysis 2: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 155 U; BOTOX 155 U vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.578, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.4, 95% CI 2-sided [-1.06 to 1.90], Standard Error of Mean 0.75 — LS Mean Difference = BOTOX 155 U - Placebo

8. Secondary Outcome: Change From Baseline in the Total 6-item Headache Impact Test (HIT-6) Score Across Months 5 and 6
Description: The HIT-6 is a 6-item assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home and in social situations. It assesses the effect that headaches have on normal daily life and the subject's ability to function. Responses are based on frequency using a 5-point scale ranging from "never" to "always." The HIT-6 total score, which ranges from 36 to 78, is the sum of the responses, each of which is assigned a score ranging from 6 points (never) to 13 points (always). The Total 6-item Headache Impact Test (HIT-6) score across Months 5 and 6 is calculated by taking the 2-month average of total 6-item Headache Impact Test (HIT-6) scores over Months 5 and 6. Negative changes from Baseline in the HIT-6 score indicate improvement.
Time Frame: Baseline, Months 5-6
Population: Intent-to-Treat Population (as Randomized); data used are "observed data" (without imputation for missing values)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U
Number analyzed (Participants) | 228 | 238 | 229
units on a scale | -6.2 [-7.26 to -5.08] | -6.9 [-7.94 to -5.77] | -6.5 [-7.62 to -5.45]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 195 U; BOTOX 195 U vs Placebo; Test type: Superiority — P-value/95% CI are obtained from a mixed-effects model for repeated measures (MMRM) analysis for primary analysis of the 2 visits across Months 5 and 6. Tx (BOTOX 195 U, BOTOX 155 U, placebo), month (Months 1-6), country, strata of previous exposure to migraine prophylactic treatment, and Tx group-by-month interaction as fixed effects, with the Baseline total HIT-6 score as a covariate, included as a continuous variable. Subject and residual errors are random effects; p = 0.589, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.4, 95% CI 2-sided [-1.69 to 0.96], Standard Error of Mean 0.68 — LS Mean Difference = BOTOX 195 U - Placebo
Statistical Analysis 2: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: BOTOX 155 U; BOTOX 155 U vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.310, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.7, 95% CI 2-sided [-2.00 to 0.64], Standard Error of Mean 0.67 — LS Mean Difference = BOTOX 155 U - Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from time informed consent was signed to end of the study. Median time on follow-up was 30 days in the Screening/Baseline Phase; 168 days in the Double-Blind Phase; and 169 days in the Open-Label Phase.
Description: Participants were analyzed according to the study treatment that they actually received at the first injection cycle on Day 1. For safety analysis, there was 1 participant who belonged to a different treatment group than assigned by randomization (BOTOX 195 U instead of BOTOX 155 U).
Arm/Group | Screening/Baseline Phase | Double-Blind Phase: Placebo | Double-Blind Phase: BOTOX 155 U | Double-Blind Phase: BOTOX 195 U | Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U | Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U
All-Cause Mortality (participants affected / at risk) | 0/775 | 0/257 | 0/256 | 1/262 | 0/217 | 0/227 | 1/223
Serious Adverse Events (participants affected / at risk) | 2/775 | 6/257 | 3/256 | 6/262 | 2/217 | 1/227 | 1/223
Other Adverse Events (participants affected / at risk) | 14/775 | 21/257 | 35/256 | 22/262 | 19/217 | 18/227 | 14/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening/Baseline Phase (N=775) | Double-Blind Phase: Placebo (N=257) | Double-Blind Phase: BOTOX 155 U (N=256) | Double-Blind Phase: BOTOX 195 U (N=262) | Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U (N=217) | Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U (N=227) | Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U (N=223)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PORTOSPLENOMESENTERIC VENOUS THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIPOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MIGRAINE WITH AURA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LABILE BLOOD PRESSURE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening/Baseline Phase (N=775) | Double-Blind Phase: Placebo (N=257) | Double-Blind Phase: BOTOX 155 U (N=256) | Double-Blind Phase: BOTOX 195 U (N=262) | Double-Blind Phase: Placebo/Open-Label Phase: BOTOX 195 U (N=217) | Double-Blind Phase: BOTOX 155 U/Open-Label Phase: BOTOX 195 U (N=227) | Double-Blind Phase: BOTOX 195 U/Open-Label Phase: BOTOX 195 U (N=223)
COVID-19 (Infections and infestations) | 4 (4) | 9 (9) | 16 (16) | 8 (8) | 12 (12) | 9 (9) | 7 (7)
NASOPHARYNGITIS (Infections and infestations) | 10 (10) | 14 (15) | 23 (26) | 15 (18) | 7 (10) | 10 (12) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT05028569/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT05028569/SAP_001.pdf